CLINICAL TRIAL: NCT05350176
Title: Effects of Probiotic Supplementation on Sport Performance and Gut Damage in CrossFit
Brief Title: Probiotic Supplementation in Sport Performance and Gut Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Asier Santibañez, MsC, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Lact.Bas
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Sport Performance; Gut Damage
Keywords: Probiotic; Gut damage; Sport performance
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Probiotic intake containing 10 billions of Colony Forming Units of Lactobacillus plantarum (1 capsule per day)
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Placebo intake. Placebo capsules will contain dextrose (1 capsule per day)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic capsules will be composed of 10 billion CFU of Lactobacillus plantarum.
  Arms: Experimental group
Dietary Supplement: Placebo — Capsules containing dextrose (1 capsule per day)
  Arms: Placebo group

SUMMARY:
This study will be performed with the aim to evaluate the effects of probiotic supplementation on sport performance and gut damage. Participants will be divided into two groups, placebo and experimental group. With the purpose to assess the effects of probiotics on the gut damage, a strenuous exercise session will be performed, and then blood samples will be taken to observe the variation of the selected intestinal damage marker. 24 hours after this strenuous session, performance tests will be performed. After the 4 weeks of supplementation, the same procedure will be followed to evaluate the effect of probiotics.

DETAILED DESCRIPTION:
One week before the initiation of the study participants will be required to avoid consuming drugs, alcohol, cigarettes, probiotics, and any other food or liquid which could modify gut microbiota composition. For the baseline values, height, weight and sports performance test, of the participants will be collected. The same day, a strenuous exercise session will be performed in order to observe the variation of the intestinal damage marker (blood sample extraction just after finishing the strenous exercise session). 24 hours after that session sport performance tests will be conducted. Participants will then be randomly divided into two groups, one of which will take one probiotic capsule per day containing 10 billion colony-forming units (CFU) of Lactobacillus plantarum, and the other group will take one placebo capsule per day consisting of dextrose. The supplementation period will last 4 weeks.

After the supplementation period, the same process will be followed, with the same strenuous exercise session and immediate blood sampling to determine the effects of probiotics on the intestinal damage caused by exercise. 24 hours later, performance tests will be conducted to assess the effects of probiotics on sport performance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* No injuries
* 1 year of CrossFit practicing experience

Exclusion Criteria:

* Drug, alcohol, cigarettes, probiotic intake
* Injuries

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Intestinal-fatty acid-binding protein | 0-10 minutes after strenuous exercise blood samples will be extracted
  Gut damage marker
Counter movement jump test | 24 hours after strenuous training session. First test to be performed
  Jumping test
Running Based Anaerobic Sprint Test | 24 hours after strenuous training session. Second test to be performed
  Running test
YO YO Intermittent Recovery Level test 1 | 24 hours after strenuous training session. Third test to be performed
  aerobic test

CONTACTS AND LOCATIONS:
Overall Officials: Asier Santibañez, MsC, Principal Investigator — University of the Basque Country (UPV/EHU)
Locations (1):
- CrossFit Bikain, Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: No